CLINICAL TRIAL: NCT04248673
Title: Düsseldorf Bread Study on Health Effects of Bread.
Brief Title: Düsseldorf Bread Study
Acronym: DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: Bakery Hinkel (Unknown)
Responsible Party: Principal Investigator, Stephan Martin, director, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Bread study
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbohydrate rich bread (Placebo Comparator)
  Interventions: Other: carbohydrate rich bread
- carbohydrate reduced bread (Experimental)
  Interventions: Other: carbohydrate reduced bread

INTERVENTIONS:
Other: carbohydrate reduced bread — Consumption of carbohydrate reduced bread for three months.
  Arms: carbohydrate reduced bread
Other: carbohydrate rich bread — Consumption of carbohydrate rich bread for three months.
  Arms: carbohydrate rich bread

SUMMARY:
The hypothesis is to be tested that eating carbohydrate-reduced bread over three months leads to a significant weight difference compared to conventional, carbohydrate-rich bread.

DETAILED DESCRIPTION:
Carbohydrate reduction is an important element for weight loss or can also be used to keep weight constant. Since the majority of the carbohydrates consumed daily in industrialized countries come from bread and rolls, the present study will examine the effect of two different types of bread on the weight development of overweight bread consumers. The two types of bread differ in their carbohydrate content and the hypothesis is to be tested that eating carbohydrate-reduced bread over three months leads to a significant weight difference compared to conventional, carbohydrate-rich bread. The comparison of the two types of bread is carried out triple blinded. During two visits (before and after the bread consumption phase), the health status is determined with physical parameters and laboratory parameters from a blood test. The primary endpoint is body weight. Overall, this study will for the first time allow extensive statements to be made on the health value of the three-month consumption of two different types of bread.

ELIGIBILITY:
Inclusion Criteria:

- body mass index of at least 27 kg/m2

Exclusion Criteria:

* serious illness with hospitalization in the last 3 months
* Changes in body weight (estimated weekly average) by more than 2 kg in the past 4 weeks
* Non-smoking status for less than 3 months
* Change of smoking habits planned during the study
* acute diseases such as respiratory or gastrointestinal infections
* Chronic diseases, e.g. Tumor diseases, chronic obstructive pulmonary disease (COPD), asthma, dementia, intestinal diseases, diabetes
* regular use of medication (except contraceptives) such as Lipid lowering, blood pressure lowering, weight-regulating medication, aspirin
* no contraception in women of childbearing age or breastfeeding a child
* high sporting activity (≥ 1 hour per day)
* planned absence of> 7 days during the intervention phase

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
body weight | 3 months
  change of body weight in kg

SECONDARY OUTCOMES:
body mass index | 3 months
  change of body mass index in kg/m*m (body weight and height will be combined to report body mass index)
waist circumference | 3 months
  change of weight circumference in cm
waist-to-height-index | 3 months
  change of waist-to-height-index (waist circumference and height will be combined to report waist-to-height-index)
hip circumference | 3 months
  change of hip circumference in cm
blood pressure | 3 months
  change of blood pressure in mmHg
triglycerides | 3 months
  change of triglycerides in mg/dl
total cholesterol | 3 months
  change of total cholesterol in mg/dl
high-density lipoprotein (HDL) cholesterol | 3 months
  change of high-density lipoprotein (HDL) cholesterol in mg/dl
low-density lipoprotein (HDL) cholesterol | 3 months
  change of low-density lipoprotein (HDL) cholesterol in mg/dl
hemoglobin A1c (HbA1C) | 3 months
  change of hemoglobin A1c (HbA1C) in %
fasting blood glucose | 3 months
  change of fasting blood glucose in mg/dl
fasting blood insulin | 3 months
  change of fasting blood insulin µU/ml
homeostasis model assessment of insulin resistance (HOMA-IR) | 3 months
  change of homeostasis model assessment of insulin resistance (HOMA-IR) (fasting blood glucose and fasting blood insulin will be combined to report HOMA-IR)
height | at baseline
  height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- West German Centre of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No